CLINICAL TRIAL: NCT00946777
Title: Barrier Function Measurement in Dry Eye Patients After Using Systane Ultra for 30 Days
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-09-04
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: Dry Eye Signs; barrier function
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Systane® Ultra (Experimental)
  Interventions: Other: Systane® Ultra

INTERVENTIONS:
Other: Systane® Ultra — Systane® Ultra 1-2 drops, 4 times per day for 30 days

SUMMARY:
The primary objective is to determine if there is a correlation between reductions in corneal staining and improvements in corneal barrier function.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have moderate corneal staining and exhibit a need to use artificial tears.

Exclusion Criteria:

* Patients can not participate in any other ophthalmic drug or device clinical trial within 30 days of the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline of corneal fluorescein | 30 days

SECONDARY OUTCOMES:
Adverse event occurence | 30 Days

REFERENCES:
- [Result] Fernandez KB, Epstein SP, Raynor GS, Sheyman AT, Massingale ML, Dentone PG, Landegger LD, Asbell PA. Modulation of HLA-DR in dry eye patients following 30 days of treatment with a lubricant eyedrop solution. Clin Ophthalmol. 2015 Jun 24;9:1137-45. doi: 10.2147/OPTH.S81355. eCollection 2015. PMID 26170605